CLINICAL TRIAL: NCT00447824
Title: Pain Detection and Interception in Neonates During Blood Sampling
Brief Title: Pain Detection and Interception in Neonates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: Helse sor (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-06471a
Record Dates: First submitted 2007-03-13; First posted 2007-03-15 (Estimated); Last update posted 2007-03-15 (Estimated); Status verified 2007-03

CONDITIONS: Pain Detection; Pain Intervention
Keywords: Pain; Neonates; NIDCAP; Venous; Capillary
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Introduction of better conditions during blood sampling

SUMMARY:
Hypothesis:

1. May the introduction of NIDCAP during blood sample reduced pain in neonates during blood sample
2. Compare the effect of venous and capillary blood sample method

DETAILED DESCRIPTION:
introducing the: Newborn Individualized Developmental Care and Assessment Program

ELIGIBILITY:
Inclusion Criteria:

* Born gestation age 31-36

Exclusion Criteria:

* Infection, respiratory distress

Ages: 31 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160
Dates: Start 2007-03; Study Completion 2009-11

PRIMARY OUTCOMES:
value of Premature Infant Pain Profile
Heart rate
Saturation
Skin conductance changes

CONTACTS AND LOCATIONS:
Overall Officials: Knut G Hernes, Dr, Study Chair
Locations (1):
- Sorlandet Hospital SSHF, Kristiansand, Vest Agder, Norway